CLINICAL TRIAL: NCT00783575
Title: Genetic Markers as Predictors of Phenotypes in Pediatric Onset Crohn's Disease
Status: Withdrawn | Type: Observational
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: CHW 02/142
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Crohn's disease; Ulcerative colitis; Inflammatory bowel disease; NOD2,CARD 15 mutations
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extraction, serology
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease: Crohn's disease (CD) and ulcerative colitis (UC), collectively known as inflammatory bowel disease (IBD) are chronic, life-long, destructive inflammatory conditions of the gastrointestinal tract.

SUMMARY:
The purpose of this study is to look for the NOD2 gene in children with Inflammatory Bowel Disease (IBD) and their parents. We hope to understand this NOD2 gene better by determining whether children that have IBD have the NOD2 gene. In those with the NOD2 gene, we want to see if the type of gene abnormality predicts the nature of their disease and if the genetic information helps doctors decide what therapies and/or treatments to use for their patients. We also hope to explore the relationships between known serologic markers of IBD (ASCA, pANCA, ompC) and the clinical characteristics and course of children with IBD.

About 1500 children and as many of their parents as possible will take part in this study. Children who are newly diagnosed with IBD as well as children that are being seen in the Children's Health System are eligible to participate in this study. We are looking for children 18 years old or younger to participate. If possible, we would also like both parents of the child to participate.

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC), collectively known as inflammatory bowel disease (IBD) are chronic, life-long, destructive inflammatory conditions of the gastrointestinal tract. IBD onset can occur at any age but the highest incidence occurs in late childhood, adolescence and young adulthood. The incidence of IBD in children and adolescents has significantly increased over the last 40 years. The precise factors underlying IBD pathogenesis are not yet defined but may involve persistent bacterial infection, a defective mucosal barrier, or an imbalance in the regulation of the immune response. Epidemiologic studies from adult populations have identified a significant genetic contribution to the etiology of CD, but simple Mendelian models of IBD inheritance are not supported by segregation analysis. Taken together, these observations support a complex immunogenetic model of IBD whereby genetically susceptible individuals harbor an aberrant response to yet-unidentified environmental influences. Attempts to localize IBD susceptibility genes through genome-wide linkage studies have identified putative loci on chromosome 16. Recently 3 groups of investigators have shown that sequence variations within the NOD2 gene (MIM 605956) on chromosome 16q12 were strongly associated with susceptibility to CD. Attempts to link NOD2 mutations with disease phenotype have recently identified an association between ileal specific-disease and patients with NOD2/ CARD 15 mutations. This initial association between genotype and phenotype suggests that genetic factors influence disease location. At this time the frequency of NOD2 gene mutations in a population based sample, specifically in a cohort of newly diagnosed patients is not known. In addition, all attempts to correlate genotype with CD phenotype have been performed in adults, and no data has been generated in children. Identification of these mutations in children will be of particular interest, as the presentation of initial disease will manifest disease in its "purest" form, where the long duration of chronic inflammation typically seen in adult patients will not have exerted influence on disease phenotype (i.e. stricture formation secondary to longstanding, poorly controlled inflammation). Thus, genotype/phenotype correlation in children in a prospective fashion will function to characterize NOD2/ CARD15 mutations in a general population, and will also begin the evaluation of disease progression and prediction of disease severity and behaviour over time, with the starting point being the time of diagnosis. This will have obvious clinical and therapeutic implications, and will begin the process of linking disease genotype to optimal therapy. Therefore, our central hypothesis: Identification of NOD2/ CARD 15 mutations in newly diagnosed CD children will predict disease location, disease behaviour and will identify optimal approaches to therapy. This will be tested by the following three Specific Aims.

1. Genotype a cohort of WI IBD children for 4 NOD2 / CARD 15 mutations.
2. Statistical analysis of phenotype and genotype correlation in a cohort of WI pediatric IBD alliance children with or without a family history of IBD.

The Wisconsin pediatric IBD alliance was formed in January of 2000 to track all new diagnoses of IBD occurring in children younger than age 18. This clinical consortium has successfully recruited 100% of the pediatric GI specialists within Wisconsin to prospectively record all new IBD diagnoses, in order to obtain a population based incidence of CD and UC within the U.S. Between 1/1/00 and 12/31/01, we have identified 192 new cases of IBD within the state. Sixty-five percent of these children were from Southeast Wisconsin, and were diagnosed at Children's Hospital of Wisconsin. In addition to these newly diagnosed children, a cohort of 294 additional pediatric IBD children followed at the Children's Hospital of Wisconsin will serve as a reference population. The focus of this proposal will be to correlate genetic influence on the clinical disease course and behavior using a molecular classification of pediatric CD children in a population based pediatric cohort. This DDC grant will allow the PI and the co-investigator to generate sufficient preliminary data in the under-researched area of pediatric CD and to continue this investigation for support from national foundations (CCFA) and /or the NIH.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Inflammatory Bowel Disease (Crohn's Disease, ulcerative colitis or indeterminate colitis).

Exclusion Criteria:

* Diagnosis during non-pediatric age.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from Southeast Wisconsin diagnosed with Inflammatory Bowel Disease at Children's Hospital of Wisconsin and their biological parents.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2002-10; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Genotype a cohort of IBD children for 4 NOD2/CARD15 mutations. | Study completion

SECONDARY OUTCOMES:
Statistical analysis of phenotype and genotype correlation in a cohort of pediatric Inflammatory Bowel Disease children with or without a family history of Inflammatory Bowel Disease | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stephens, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Sawczenko A, Sandhu BK, Logan RF, Jenkins H, Taylor CJ, Mian S, Lynn R. Prospective survey of childhood inflammatory bowel disease in the British Isles. Lancet. 2001 Apr 7;357(9262):1093-4. doi: 10.1016/s0140-6736(00)04309-9. PMID 11297962
- [Background] Orchard TR, Satsangi J, Van Heel D, Jewell DP. Genetics of inflammatory bowel disease: a reappraisal. Scand J Immunol. 2000 Jan;51(1):10-7. doi: 10.1046/j.1365-3083.2000.00656.x. PMID 10632970
- [Background] Ahmad T, Armuzzi A, Bunce M, Mulcahy-Hawes K, Marshall SE, Orchard TR, Crawshaw J, Large O, de Silva A, Cook JT, Barnardo M, Cullen S, Welsh KI, Jewell DP. The molecular classification of the clinical manifestations of Crohn's disease. Gastroenterology. 2002 Apr;122(4):854-66. doi: 10.1053/gast.2002.32413. PMID 11910336
- [Background] Podolsky DK. Inflammatory bowel disease (1). N Engl J Med. 1991 Sep 26;325(13):928-37. doi: 10.1056/NEJM199109263251306. No abstract available. PMID 1881418
- [Background] Podolsky DK. Inflammatory bowel disease (2). N Engl J Med. 1991 Oct 3;325(14):1008-16. doi: 10.1056/NEJM199110033251406. No abstract available. PMID 1886623
- [Background] Hugot JP, Laurent-Puig P, Gower-Rousseau C, Olson JM, Lee JC, Beaugerie L, Naom I, Dupas JL, Van Gossum A, Orholm M, Bonaiti-Pellie C, Weissenbach J, Mathew CG, Lennard-Jones JE, Cortot A, Colombel JF, Thomas G. Mapping of a susceptibility locus for Crohn's disease on chromosome 16. Nature. 1996 Feb 29;379(6568):821-3. doi: 10.1038/379821a0. PMID 8587604
- [Background] Hampe, J. and S. Schrieber, A genome-wide search identies potential susceptibility loci for Crohn's disease. Am J Hum Genet, 1999. 64: p. 808-16.
- [Background] Hugot JP, Chamaillard M, Zouali H, Lesage S, Cezard JP, Belaiche J, Almer S, Tysk C, O'Morain CA, Gassull M, Binder V, Finkel Y, Cortot A, Modigliani R, Laurent-Puig P, Gower-Rousseau C, Macry J, Colombel JF, Sahbatou M, Thomas G. Association of NOD2 leucine-rich repeat variants with susceptibility to Crohn's disease. Nature. 2001 May 31;411(6837):599-603. doi: 10.1038/35079107. PMID 11385576
- [Background] Ogura Y, Bonen DK, Inohara N, Nicolae DL, Chen FF, Ramos R, Britton H, Moran T, Karaliuskas R, Duerr RH, Achkar JP, Brant SR, Bayless TM, Kirschner BS, Hanauer SB, Nunez G, Cho JH. A frameshift mutation in NOD2 associated with susceptibility to Crohn's disease. Nature. 2001 May 31;411(6837):603-6. doi: 10.1038/35079114. PMID 11385577
- [Background] Calkins, B.M., Inflammatory Bowel Diseases, in Digestive Diseases in the United States: Epidemiology and Impact, J.E. Everhart, Editor. 1994, U.S. Government Printing Office: Washington D.C. p. 509-550.
- [Background] Sandborn WJ. A review of immune modifier therapy for inflammatory bowel disease: azathioprine, 6-mercaptopurine, cyclosporine, and methotrexate. Am J Gastroenterol. 1996 Mar;91(3):423-33. No abstract available. PMID 8633486
- [Background] D'Haens GR, Gasparaitis AE, Hanauer SB. Duration of recurrent ileitis after ileocolonic resection correlates with presurgical extent of Crohn's disease. Gut. 1995 May;36(5):715-7. doi: 10.1136/gut.36.5.715. PMID 7797122
- [Background] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078
- [Background] Barton JR, Gillon S, Ferguson A. Incidence of inflammatory bowel disease in Scottish children between 1968 and 1983; marginal fall in ulcerative colitis, three-fold rise in Crohn's disease. Gut. 1989 May;30(5):618-22. doi: 10.1136/gut.30.5.618. PMID 2786488
- [Background] Cosgrove M, Al-Atia RF, Jenkins HR. The epidemiology of paediatric inflammatory bowel disease. Arch Dis Child. 1996 May;74(5):460-1. doi: 10.1136/adc.74.5.460. PMID 8669968
- [Background] Armitage E, Drummond H, Ghosh S, Ferguson A. Incidence of juvenile-onset Crohn's disease in Scotland. Lancet. 1999 May 1;353(9163):1496-7. doi: 10.1016/S0140-6736(99)00333-5. No abstract available. PMID 10232323
- [Background] Satsangi J, Parkes M, Louis E, Hashimoto L, Kato N, Welsh K, Terwilliger JD, Lathrop GM, Bell JI, Jewell DP. Two stage genome-wide search in inflammatory bowel disease provides evidence for susceptibility loci on chromosomes 3, 7 and 12. Nat Genet. 1996 Oct;14(2):199-202. doi: 10.1038/ng1096-199. PMID 8841195
- [Background] Forabosco P, Collins A, Latiano A, Annese V, Clementi M, Andriulli A, Fortina P, Devoto M, Morton NE. Combined segregation and linkage analysis of inflammatory bowel disease in the IBD1 region using severity to characterise Crohn's disease and ulcerative colitis. On behalf of the GISC. Eur J Hum Genet. 2000 Nov;8(11):846-52. doi: 10.1038/sj.ejhg.5200542. PMID 11093274
- [Background] Orholm M, Iselius L, Sorensen TI, Munkholm P, Langholz E, Binder V. Investigation of inheritance of chronic inflammatory bowel diseases by complex segregation analysis. BMJ. 1993 Jan 2;306(6869):20-4. doi: 10.1136/bmj.306.6869.20. PMID 8435571
- [Background] Monsen U, Iselius L, Johansson C, Hellers G. Evidence for a major additive gene in ulcerative colitis. Clin Genet. 1989 Dec;36(6):411-4. PMID 2591066
- [Background] Spielman RS, Ewens WJ. The TDT and other family-based tests for linkage disequilibrium and association. Am J Hum Genet. 1996 Nov;59(5):983-9. No abstract available. PMID 8900224
- [Background] Cho JH, Nicolae DL, Gold LH, Fields CT, LaBuda MC, Rohal PM, Pickles MR, Qin L, Fu Y, Mann JS, Kirschner BS, Jabs EW, Weber J, Hanauer SB, Bayless TM, Brant SR. Identification of novel susceptibility loci for inflammatory bowel disease on chromosomes 1p, 3q, and 4q: evidence for epistasis between 1p and IBD1. Proc Natl Acad Sci U S A. 1998 Jun 23;95(13):7502-7. doi: 10.1073/pnas.95.13.7502. PMID 9636179
- [Background] Rioux JD, Silverberg MS, Daly MJ, Steinhart AH, McLeod RS, Griffiths AM, Green T, Brettin TS, Stone V, Bull SB, Bitton A, Williams CN, Greenberg GR, Cohen Z, Lander ES, Hudson TJ, Siminovitch KA. Genomewide search in Canadian families with inflammatory bowel disease reveals two novel susceptibility loci. Am J Hum Genet. 2000 Jun;66(6):1863-70. doi: 10.1086/302913. Epub 2000 Apr 21. PMID 10777714
- [Background] Rioux JD, Daly MJ, Silverberg MS, Lindblad K, Steinhart H, Cohen Z, Delmonte T, Kocher K, Miller K, Guschwan S, Kulbokas EJ, O'Leary S, Winchester E, Dewar K, Green T, Stone V, Chow C, Cohen A, Langelier D, Lapointe G, Gaudet D, Faith J, Branco N, Bull SB, McLeod RS, Griffiths AM, Bitton A, Greenberg GR, Lander ES, Siminovitch KA, Hudson TJ. Genetic variation in the 5q31 cytokine gene cluster confers susceptibility to Crohn disease. Nat Genet. 2001 Oct;29(2):223-8. doi: 10.1038/ng1001-223. PMID 11586304
- [Background] Lesage S, Zouali H, Cezard JP, Colombel JF, Belaiche J, Almer S, Tysk C, O'Morain C, Gassull M, Binder V, Finkel Y, Modigliani R, Gower-Rousseau C, Macry J, Merlin F, Chamaillard M, Jannot AS, Thomas G, Hugot JP; EPWG-IBD Group; EPIMAD Group; GETAID Group. CARD15/NOD2 mutational analysis and genotype-phenotype correlation in 612 patients with inflammatory bowel disease. Am J Hum Genet. 2002 Apr;70(4):845-57. doi: 10.1086/339432. Epub 2002 Mar 1. PMID 11875755